CLINICAL TRIAL: NCT02093338
Title: Study of Intervention Nutritional, Multicenter, Randomized, Blind, Parallel Group to Evaluate the Efficacy of Lactobacillus Fermentum CECT5716 to Reduce the Load Bacterial in Potential Pathogens in Milk of Mothers With Breast Pain
Brief Title: L.Fermentum CECT5716 in Treatment of Breast Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Biosearch S.A. (Industry)
Collaborators: Junta de Andalucia (Other Government); Statistical analysis: SEPLIN Soluciones Estadísticas (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: P025
Record Dates: First submitted 2013-07-18; First posted 2014-03-21 (Estimated); Last update posted 2014-03-21 (Estimated); Status verified 2014-03

CONDITIONS: Breast Pain
Keywords: breast pain; probiotic; mastitis; lactobacillus fermentun; Staphylococcus
MeSH Terms: conditions — Mastodynia; Mastitis

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- fermentum 3x (Experimental): Lactobacillus fermentum CECT5716 at 3x10e9 cfu/day
  Interventions: Dietary Supplement: Lactobacillus fermentum CECT5716
- fermentum 6x (Experimental): Lactobacillus fermentum CECT5716 at 6x10e9cfu/day
  Interventions: Dietary Supplement: Lactobacillus fermentum CECT5716
- fermentum 9x (Experimental): Lactobacillus fermentum CECT5716 at 9x10e9cfu/day
  Interventions: Dietary Supplement: Lactobacillus fermentum CECT5716
- maltodextrin (Placebo Comparator): maltodextrin
  Interventions: Other: Placebo Comparator: maltodextrin

INTERVENTIONS:
Dietary Supplement: Lactobacillus fermentum CECT5716
  Arms: fermentum 3x; fermentum 6x; fermentum 9x
Other: Placebo Comparator: maltodextrin — Placebo
  Arms: maltodextrin

SUMMARY:
The main objective of this intervention study is to evaluate the efficacy of Lactobacillus fermentum CECT5716 to reduce the presence in the milk of genera Staphylococcus and Streptococcus as risk factors for mastitis in women with breast pain

DETAILED DESCRIPTION:
1. Type of study Nutritional intervention study, multicenter, randomized, blinded, parallel group included 25 women per group

   * Group 1: 3x109 cfu / day (n = 25)
   * Group 2: 6x109 cfu / day (n = 25)
   * Group 3: 9x109 cfu / day (n = 25)
   * Group 4: placebo (n = 25)
2. Statistical calculation of sample size. The calculation of sample size was calculated by the company SEPLIN Solutions Statistics. The primary endpoint was the bacterial count of in milk. The sample size obtained to observe a difference of 1 log10, with a power of 0.80 and a significance level of 0.05 was 20 volunteers per group.
3. Randomization Randomization was performed using a list of random numbers generated by computer. Subjects will be randomized in a strictly sequential.

   If a subject is removed from the test, the number that was assigned randomization not be reused again.
4. Overall design and outline of the study At visit 1 we require the informed consent of the patient. It will take the milk sample, we will review the implementation of the inclusion and exclusion criteria. Be randomized and explain the treatment guidelines to be followed, the data to be collected and medical appointments that must go (2 and 3 weeks). It will complete the pain assessment questionnaire (MQP) and nutrition survey.

   On visits 2, 3 and 4 corresponding to 1, 2 and 3 weeks of intervention will collect milk sample pain assessment survey and nutrition survey.

   Milk samples (5 mL) were collected aseptically in sterile tubes to be frozen immediately until analysis to be carried out within seven days.
5. Intervention duration The intervention will last three weeks.

ELIGIBILITY:
Inclusion Criteria:

· breast-feeding women

* Swelling and / or warmth in the chest
* Chest pain
* total bacteria count in milk greater than or equal to 3 log10 colony forming units (CFU) / mL,

Exclusion Criteria:

* breast abscesses, Raynaud syndrome,
* Antibiotic treatment
* Allergic to antibiotics
* Low expectation of compliance with the study protocol.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 127 (Actual)
Dates: Start 2011-07; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Change from baseline Staphylococcus count at 3 weeks | 0, 3 weeks
  Counts of Staphylococcus in breast milk

SECONDARY OUTCOMES:
Change from baseline Streptococcus counts at 3 weeks | 0, 3 weeks
  Streptococcus counts in breast milk
Change from Breast pain score at 3 weeks | 0, 3 weeks
  evaluation of breast pain

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Miguel A Díaz López, Doctor, Principal Investigator — Gynecology Service of Virgen de las Nieves Hospital, Granada (Spain)
Locations (1):
- Hospital Virgen de las Nieves, Granada, Granada, Spain

REFERENCES:
- [Derived] Crepinsek MA, Taylor EA, Michener K, Stewart F. Interventions for preventing mastitis after childbirth. Cochrane Database Syst Rev. 2020 Sep 29;9(9):CD007239. doi: 10.1002/14651858.CD007239.pub4. PMID 32987448